CLINICAL TRIAL: NCT03184350
Title: Adjuvant Protontherapy of Cervical and Endometrial Carcinomas - A Phase-II-study
Brief Title: Adjuvant Protontherapy of Cervical and Endometrial Carcinomas
Acronym: APROVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nils Nicolay, PD Dr. Dr., senior physician, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APROVE
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Uterine Cervical Neoplasms; Endometrial Neoplasms Malignant
Keywords: cervical cancer; endometrial cancer; proton therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will receive a dose of 45-50.4 Gray in 1.8 Gray fractions 5-6 times per week using active raster-scanning pencil beam proton radiation. Platinum-based chemotherapy can be administered if indicated. For treatment planning rectum, sigma, large and small bowel, bladder and femoral heads are defined as organs at risk. The CTV is defined according to the EORTC consensus guidelines. Treatment-associated toxicity and Quality of life will be evaluated regularly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant pelvic proton radiation (Other)
  Interventions: Radiation: Adjuvant pelvic proton radiation

INTERVENTIONS:
Radiation: Adjuvant pelvic proton radiation — Patients will receive a dose of 45-50.4 Gray in 1.8 Gray fractions 5-6 times per week using active raster-scanning pencil beam proton radiation

SUMMARY:
The APROVE study is a prospective single-center single-arm phase-II study. Patients with cervical or endometrial cancer after surgical resection who have an indication for postoperative pelvic radiotherapy will be treated with proton therapy instead of the commonly used photon radiation. A total of 25 patients will be included in this trial. Patients will receive a dose of 45-50.4 Gray in 1.8 Gray fractions 5-6 times per week using active raster-scanning pencil beam proton radiation. Platinum-based chemotherapy can be administered if indicated. The primary endpoint of the study is the evaluation of safety and treatment tolerability of pelvic radiation using protons defined as the lack of any CTC AE Grade 3 or 4 toxicity. Secondary endpoints are clinical symptoms and toxicity, quality of life and progression-free survival. The aim is to explore the potential of proton therapy as a new method for adjuvant pelvic radiotherapy to decrease the dose to the bowel, rectum and bladder thus reducing acute and chronic toxicity and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical or endometrial cancer
* Indication for postoperative radiotherapy
* Karnofsky Index ≥ 70
* Age between 18 and 80 years
* Written informed consent

Exclusion Criteria:

* patient refusal or patient incapable of consent
* implanted active medical devices with no approval for ion beam radiation
* metallic implantations in the radiation field like hip prothesis
* prior pelvic irradiation
* participation in another clinical trial which might influence the results of the APROVE trial

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute treatment-associated adverse events ≥ grade 3 [Safety and Tolerability] | 3 months
  Assessment of toxicity according to the CTC AE v4.0 (Common Toxicity Criteria for adverse events)

SECONDARY OUTCOMES:
clinical symptoms according to the CTC AE v4.0. criteria | 2 years
  clinical symptoms of any grade will be assessed
Quality of life of all patients included in the study | 2 years
  assessed by the EORTC questionnaires QLQ-C30
Quality of life of cervical cancer patients included in the study | 2 years
  assessed by the EORTC questionnaires QLQ-CX24
Quality of life of endometrial cancer patients included in the study | 2 years
  assessed by the EORTC questionnaires QLQ-EN24
Progression-free survival | 2 years
  regular MRI-scans

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof.Dr.Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Department of radiation oncology, University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meixner E, Wark A, Forster T, Weykamp F, Lang K, Konig L, Lindel K, Oelmann-Avendano JT, Krisam J, Schneeweiss A, Ellerbrock M, Mielke T, Horner-Rieber J, Herfarth K, Debus J, Arians N. Health-related quality of life and patient-reported symptoms after postoperative proton beam radiotherapy of cervical and endometrial cancer: 2-year results of the prospective phase II APROVE-trial. Radiat Oncol. 2023 Jan 9;18(1):5. doi: 10.1186/s13014-023-02198-4. PMID 36624483
- [Derived] Arians N, Lindel K, Krisam J, Herfarth K, Krug D, Akbaba S, Oelmann-Avendano J, Debus J. Prospective phase-II-study evaluating postoperative radiotherapy of cervical and endometrial cancer patients using protons - the APROVE-trial. Radiat Oncol. 2017 Nov 28;12(1):188. doi: 10.1186/s13014-017-0926-5. PMID 29179751